CLINICAL TRIAL: NCT04531462
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, 52 Weeks Phase IV Trial to Evaluate Efficacy and Safety of Oral, Once Daily Empagliflozin in Elderly Japanese Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control
Brief Title: A Study to Test How Well Empagliflozin Works in Japanese People With Type 2 Diabetes Who Are Older Than 65 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245-0218
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 10 mg (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Arms: Empagliflozin 10 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy of empagliflozin 10 mg after 52 weeks compared to placebo in elderly patients with Type 2 diabetes mellitus (T2DM) and to explore if empagliflozin has any impact on patient physical condition compared to placebo in elderly patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Japanese (defined as patient has parents who are Japanese) patients with diagnosis of Type 2 diabetes mellitus (T2DM) prior to informed consent
* Glycated hemoglobin (HbA1c) ≥7.0% and ≤10.0% for patients at Visit 1 (screening). If the patient is on treatment with oral antidiabetic drug(s) potentially associated with severe hypoglycaemia (e.g., sulfonylurea or glinides), the following HbA1c value is used as criterion

  * HbA1c ≥7.5% and ≤10.0% for age ≥65 and <75
  * HbA1c ≥8.0% and ≤10.0% for age ≥75
* Patients on diet and exercise regimen who are drug-naïve (drug-naïve is defined as no antidiabetic drugs for at least 12 weeks prior to informed consent) or on treatment with any oral antidiabetic drug (OAD) other than Glucagon-Like Peptide-1 (GLP-1) agonists and Sodium-glucose cotransporter 2 (SGLT-2) inhibitor. Antidiabetic therapy has to be unchanged for 12 weeks prior to randomisation (any thiazolidinedione therapy has to be unchanged for at least 18 weeks prior to informed consent).
* Age ≥65 years at informed consent
* BMI ≥22 kg/m2 at Visit 1 (screening)
* Male or post-menopausal (a point in time 12 months after a woman's last period) female patients
* Patient signed and dated written informed consent in accordance with International Conference on Harmonization (ICH)- Good Clinical Practice (GCP) and local legislation prior to admission to the Trial

Exclusion Criteria:

* Uncontrolled hyperglycaemia with a fasting glucose level >200 milligram per deciliter (mg/dL) (>11.1 millimol per Liter (mmol/L)) during run-in period
* Treatment with insulin within 12 weeks prior to informed consent
* Impaired cognitive ability as supported by Mini mental state examination (MMSE-J, defined as ≤23) and verified by the investigator at screening
* Acute coronary syndrome (ST-elevation myocardial infarction [STEMI], non-STEMI, and unstable angina pectoris), stroke or transient ischemic attack within 12 weeks prior to informed consent
* Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT = serum glutamic-pyruvic transaminase [SGPT]), aspartate aminotransferase (AST = serum glutamic-oxaloacetic transaminase[SGOT]), or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN) as determined during screening and run-in period
* Impaired renal function, defined as Estimated glomerular filtration rate (eGFR) <45 milliliter per minute per 1.73 square meter (mL/min/1.73 m2, severe renal impairment, Modification of Diet in Renal Disease (MDRD) formula) as determined during screening and run-in period
* Low grip strength defined as <28 kilogram (kg) for male or as <18 kg for female at screening
* Short length of calf circumference defined as <34 centimeter (cm) for male or 33 cm for female at screening
* further exclusion criteria apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Meitetsu Hospital, Aichi, Nagoya
  - Chubu Rosai Hospital, Aichi, Nagoya
  - Daido Hospital, Aichi, Nagoya
  - Seino Internal Medicine Clinic, Fukushima, Koriyama
  - Gifu University Hospital, Gifu, Gifu
  - Watanabe Clinic, Hyogo, Nishinomiya
  - Institute Medical Corporation Hitomikai Motomachi Takatsuka Naika Clinic, Kanagawa, Yokohama
  - Medical Corporation KEISEIKAI Kajiyama Clinic, Kyoto, Kyoto
  - Medical Corporation Hayashi Katagihara Clinic, Kyoto, Kyoto
  - Iryouhouijneiwakai Minamiakatsuka Clinic, Mito, Ibaraki
  - Moriya Keiyu Hospital, Moriya, Ibaraki
  - North Alps Medical Center Azumi Hospital, Nagano, Kitaazumi-gun
  - Asama Nanroku Komoro Medical Center, Nagano, Komoro
  - Koshigaya Municipal Hospital, Saitama, Koshigaya
  - Dojinkinenkai Meiwa Hospital, Tokyo, Chiyoda-ku
  - Tokyo Asbo Clinic, Tokyo, Chuo-ku
  - Shinagawa East one Medical Clinic, Tokyo, Minato-ku
  - Ikebukuro Metropolitan Clinic, Tokyo, Toshima-ku

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yabe D, Shiki K, Suzaki K, Meinicke T, Kotobuki Y, Nishida K, Clark D, Yasui A, Seino Y. Rationale and design of the EMPA-ELDERLY trial: a randomised, double-blind, placebo-controlled, 52-week clinical trial of the efficacy and safety of the sodium-glucose cotransporter-2 inhibitor empagliflozin in elderly Japanese patients with type 2 diabetes. BMJ Open. 2021 Apr 7;11(4):e045844. doi: 10.1136/bmjopen-2020-045844. PMID 33827843
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomised, double-blind, placebo-controlled, parallel group, multicentre trial compared 10 mg empagliflozin with placebo after 52 weeks in elderly Japanese patients with Type 2 diabetes mellitus (T2DM) and insufficient glycaemic control.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Type 2 diabetes mellitus (T2DM) Japanese patients older than 65 years administered orally once daily one film-coated tablet of placebo matching empagliflozin in addition to the standard of care treatment
- Empagliflozin 10 mg: Type 2 diabetes mellitus (T2DM) Japanese patients older than 65 years administered orally once daily one film-coated tablet 10 milligram (mg) of empagliflozin in addition to the standard of care treatment.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg
Started | 64 | 65
Completed | 58 | 61
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): This set included all patients randomised, treated with at least one dose of trial medication, and with a baseline and at least one on-treatment glycated haemoglobin (HbA1c) value.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (5.1) | 74.2 (4.9) | 74.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 44 | 48 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 63 | 64 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 64 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Percentage of glycated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycated haemoglobin] — Percentage of glycated haemoglobin (HbA1c) at baseline.
  Percentage of glycated haemoglobin | 7.6 (0.5) | 7.6 (0.5) | 7.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline After 52 Weeks of Treatment
Description: Change in glycated hemoglobin (HbA1c) (in units of %) from baseline after 52 weeks of treatment was modelled using a restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) which included fixed classification effects for treatment, gender, baseline renal function, visit and visit-by-treatment interaction, and a linear covariate for baseline HbA1c and age. The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.The Least Squares Mean (Standard Error) after 52 weeks of treatment is reported.
Time Frame: Change in HbA1c from baseline after 52 weeks of treatment was calculated using the MMRM model which is a longitudinal analyses and it incorporates HbA1c values from baseline and after 4 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks of treatment.
Population: Full Analysis Set (Observed cases): This set included all patients randomised, treated with at least one dose of trial medication, and with a baseline and at least one on-treatment HbA1c value. Only the available data that were observed while the patients were on treatment were analysed.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 62 | 64
percentage of glycated hemoglobin | -0.12 (0.08) | -0.69 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) which included fixed classification effects for treatment, gender, baseline renal function, visit and visit-by-treatment interaction, and a linear covariate for baseline HbA1c and age. An unstructured covariance structure was used to model the within patient errors. The Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Test type: Superiority — Null hypothesis: Mean change from baseline in HbA1c after 52 weeks of treatment with empagliflozin 10 mg = mean change from baseline in HbA1c after 52 weeks of treatment with placebo; p < 0.0001, Mixed Model Repeated Measures (MMRM) — Threshold level for statistical significance: α = 0.05; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.78 to -0.36] — Empagliflozin 10 mg- Placebo

2. Secondary Outcome: Change of Muscle Mass From Baseline to Week 52
Description: Muscle mass was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition, and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of muscle mass from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline muscle mass, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52
Population: Treated set (Observed cases, including values after rescue (OC-IR)): All patients randomized and treated with at least one dose of trial medication. Values measured after rescue medication were also used. Patients with missing values at Week 52 or at baseline were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | -0.96 (0.36) | -1.57 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline muscle mass, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.2310, ANCOVA; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.61 to 0.39] — Empagliflozin 10 mg- Placebo

3. Secondary Outcome: Change of Body Fat Measurement From Baseline to Week 52
Description: Body fat mass was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of body fat measurement from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline body fat measurement, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | 0.08 (0.29) | -1.77 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline body fat measurement, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.84, 95% CI 2-sided [-2.65 to -1.04] — Empagliflozin 10 mg- Placebo

4. Secondary Outcome: Change of Lean Body Mass From Baseline to Week 52
Description: Lean body mass (fat-free mass) was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition, and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of lean body mass from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline lean body mass, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | -1.08 (0.27) | -1.61 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline lean body mass, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.1632, ANCOVA; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.28 to 0.22] — Empagliflozin 10 mg- Placebo

5. Secondary Outcome: Change of Total Body Water From Baseline to Week 52
Description: Total body water was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition, and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of total body water from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline total body water, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | -0.72 (0.21) | -1.35 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline total body water, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.0384, ANCOVA; Mean Difference (Net) = -0.63, 95% CI 2-sided [-1.23 to -0.03] — Empagliflozin 10 mg- Placebo

6. Secondary Outcome: Change of Bone Mineral Content From Baseline to Week 52
Description: Bone mineral content (estimated bone mass) was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition, and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of bone mineral content from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline bone mineral content, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | -0.06 (0.02) | -0.09 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline bone mineral content, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.1975, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.01] — Empagliflozin 10 mg- Placebo

7. Secondary Outcome: Change of Skeletal Muscle Index From Baseline to Week 52
Description: Skeletal muscle index is calculated by dividing the limb muscle mass (kg) by the square of the height (m2).
  The limb muscle mass was estimated via bioelectrical impedance analysis (BIA) which is a commonly used method for estimating body composition, and it assesses body composition by passing a very small current through the body and assessing differences in impedance caused by the fact that fat and lean tissues have different electrical properties. To measure the body composition the patient barefoot stood on the bench evenly on the toe and heel electrodes and held the grip on each hand.
  Change of skeletal muscle index from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline skeletal muscle index, age, baseline glycated hemoglobin (HbA1c), baseline body mass index as linear covariates and sex, treatment as fixed effects.
  "Baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram/meter^2 (kg/m^2)
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 57 | 62
kilogram/meter^2 (kg/m^2) | -0.245 (0.064) | -0.326 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) which included baseline skeletal muscle index, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.3725, ANCOVA; Mean Difference (Net) = -0.081, 95% CI 2-sided [-0.259 to 0.098] — Empagliflozin 10 mg- Placebo

8. Secondary Outcome: Change of Grip Strength From Baseline to Week 52
Description: A Smedley-type dynamometer was used to measure grip strength. The site staff instructed the patient to adjust the grip width so that the second joint of the index finger is approximately 90 degrees (almost right angle). The site staff asked the patient to be careful not to touch the body or clothes with hand while keeping arms down naturally. The site staff made sure that the patient does not wave the grip dynamometer. Grip strength was measured twice alternately left and right.
  Change of grip strength from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline grip strength, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 59 | 62
kilogram | -0.6 (0.3) | -0.9 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline grip strength, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.4208, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.1 to 0.5] — Empagliflozin 10 mg- Placebo

9. Secondary Outcome: Change of Time in the 5-time Chair Stand Test From Baseline to Week 52
Description: For the stand test patients fold their arms across their chest and try to stand up once from a chair. If patients can stand from a chair, they repeat same action five times. It is measured the time required to perform five rise from a chair to an upright position as fast as possible without the use of arms.
  Change of time in the 5-time chair stand test from baseline to Week 52 was modelled using an Analysis of Covariance (ANCOVA) which included baseline 5-time chair stand test, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects.
  The term "baseline" refers to the last observed measurement prior to the administration of any randomised trial medication.
Time Frame: At baseline and at Week 52.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 58 | 62
seconds | -0.9 (0.3) | -0.9 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Analysis of Covariance (ANCOVA) included baseline 5-time chair stand test, age, baseline glycated hemoglobin (HbA1c), baseline body mass index (BMI) as linear covariates and sex, treatment as fixed effects; Test type: Other; p = 0.9267, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.0 to 0.9] — Empagliflozin 10 mg- Placebo

ADVERSE EVENTS:
Time Frame: From the administration of first dose of randomised trial medication until treatment stop +7 days of residual effect period, up to 378 days.
Description: Treated set: All patients randomized and treated with at least one dose of trial medication.
Groups:
- Empagliflozin 10mg: Type 2 diabetes mellitus (T2DM) Japanese patients older than 65 years administered orally once daily one film-coated tablet 10 milligram (mg) of empagliflozin in addition to the standard of care treatment.
Arm/Group | Placebo | Empagliflozin 10mg
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 8/64 | 8/65
Other Adverse Events (participants affected / at risk) | 13/64 | 14/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | Empagliflozin 10mg (N=65)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Exfoliation glaucoma (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | Empagliflozin 10mg (N=65)
Constipation (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Pyrexia (General disorders) | 3 | 4
Nasopharyngitis (Infections and infestations) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04531462/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04531462/SAP_001.pdf